CLINICAL TRIAL: NCT05771428
Title: A Randomized, Double-blind, Placebo-controlled, Dose-finding Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of ABBV-552 in Participants With Mild Alzheimer's Disease
Brief Title: Study to Assess Adverse Events, Change in Disease Activity and How Oral ABBV-552 Capsules Moves Through the Body of Participants Aged 50 to 90 Years With Mild Alzheimer's Disease
Acronym: Abroad
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-515; 2022-501918-55-00 (Other: EU CTR)
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Alzheimer's disease (AD); Dementia; ABBV-552
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ABBV-552: 1 mg (Experimental): Participants will receive 1 mg of ABBV-552 once daily (QD) for 12 weeks.
  Interventions: Drug: ABBV-552
- ABBV-552: 5 mg (Experimental): Participants will receive 5 mg of ABBV-552 QD for 12 weeks.
  Interventions: Drug: ABBV-552
- ABBV-552: 15 mg (Experimental): Participants will receive 5 mg of ABBV-552 QD for 12 weeks.
  Interventions: Drug: ABBV-552
- Placebo (Placebo Comparator): Participants will receive placebo for ABBV-552 QD for 12 weeks.
  Interventions: Drug: Placebo for ABBV-552

INTERVENTIONS:
Drug: ABBV-552 — Oral Capsule
  Arms: ABBV-552: 1 mg; ABBV-552: 15 mg; ABBV-552: 5 mg
Drug: Placebo for ABBV-552 — Oral Capsule
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is a progressive, irreversible neurological disorder and is the most common cause of dementia in the elderly population. Clinical symptoms of the disease may begin with occasional forgetfulness such as misplacement of items, forgetting important dates or events, and may progress to noticeable memory loss, increased confusion and agitation, and eventually, loss of independence and non-responsiveness. This study will assess how safe and effective ABBV-552 is in treating symptoms of early AD. Adverse events, change in disease activity, how ABBV-552 moves through body of participants and the body response to ABBV-552 will be assessed.

ABBV-552 is an investigational drug being developed for the treatment of Alzheimer's disease (AD). Study doctors put the participants in 1 of 4 groups (3 active dose groups and a placebo group), called treatment arms. Each group receives a different treatment. There is a 1 in 4 chance that participants will be assigned to placebo. Approximately 240 participants aged 50-90 years with mild AD will be enrolled in approximately 60 sites across the world.

Participants will receive oral ABBV-552 or placebo capsules once daily for 12 weeks and followed for 30 days after the last dose of study drug.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease according to the National Institute of Aging-Alzheimer's Association (NIA-AA) (2011) criteria.
* Mini-Mental State Examination (MMSE) score of 20 to 26, a Clinical Dementia Rating (CDR) global score of 0.5 or 1.0, with a CDR memory score of 0.5 or higher, and at least 1 CDR functional domain (community affairs, home and hobbies, or personal care) score of 0.5 or higher at Screening Visit 1.

Exclusion Criteria:

- Clinically significant and/or unstable medical conditions or any other reason that the investigator determines would interfere with participation in this study (e.g., unlikely to adhere to the study or procedures, keep appointments, or is planning to relocate during the study) or would make the participant an unsuitable candidate to receive ABBV-552.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (64):
- United States (37):
  - Irvine Clinical Research /ID# 250030, Irvine, California
  - Alliance for Research Alliance for Wellness /ID# 246492, Long Beach, California
  - Wake Research - Pharmacology Research Institute (WR-PRI), LLC (Alamitos) /ID# 248891, Los Alamitos, California
  - New England Institute for Clinical Research /ID# 246488, Stamford, Connecticut
  - Vertex Research Group Inc /ID# 248295, Clermont, Florida
  - Finlay Medical Research - West Palm Beach /ID# 246970, Greenacres City, Florida
  - Velocity Clinical Research - Hallandale Beach /ID# 246896, Hallandale, Florida
  - New Life Medical Research Center - Hialeah /ID# 247536, Hialeah, Florida
  - K2 Medical Research - The Villages /ID# 250820, Lady Lake, Florida
  - Allied Biomedical Res Inst Inc /ID# 246971, Miami, Florida
  - Ivetmar Medical Group, LLC. /ID# 247670, Miami, Florida
  - New Horizon Research Center /ID# 248298, Miami, Florida
  - K2 Medical Research - Ocoee /ID# 251029, Ocoee, Florida
  - Health Synergy Clinical Research LLC /ID# 247726, Okeechobee, Florida
  - K2 Medical Research - Orlando - South Orlando Avenue /ID# 250904, Orlando, Florida
  - Combined Research Orlando Phase I-IV /ID# 247697, Orlando, Florida
  - Alzheimer's Research and Treatment Center - Stuart /ID# 246484, Stuart, Florida
  - Alzheimer's Research and Treatment Center - Wellington /ID# 246491, Wellington, Florida
  - Conquest Research /ID# 262078, Winter Park, Florida
  - Columbus Memory Center /ID# 249534, Columbus, Georgia
  - Northwest Clinical Trials /ID# 248663, Boise, Idaho
  - Indiana University Health, Inc. /ID# 248300, Fort Wayne, Indiana
  - Josephson-Wallack-Munshower Neurology - Northeast /ID# 248554, Indianapolis, Indiana
  - University of Kentucky Sanders-Brown Center on Aging /ID# 251139, Lexington, Kentucky
  - NeuroMedical Clinic of Central Louisiana /ID# 246960, Alexandria, Louisiana
  - Tandem Clinical Research, LLC /ID# 246973, Marrero, Louisiana
  - Adams Clinical /ID# 248358, Watertown, Massachusetts
  - Velocity Clinical Research, Inc /ID# 249837, Raleigh, North Carolina
  - American Clinical Research Institute (ACRI) - Beavercreek /ID# 246930, Beavercreek, Ohio
  - NeuroScience Research Center - Canton /ID# 248552, Canton, Ohio
  - Neurology Diagnostics - South /ID# 246931, Dayton, Ohio
  - Duplicate_Summit Headlands LLC /ID# 250678, Portland, Oregon
  - Vanderbilt Ingram Cancer Center /ID# 248801, Nashville, Tennessee
  - Kerwin Medical Center /ID# 248662, Dallas, Texas
  - ANESC Research LLC /ID# 246958, El Paso, Texas
  - Epic Medical Research /ID# 249141, Red Oak, Texas
  - Sentara Neurology Specialists - Norfolk /ID# 248578, Norfolk, Virginia
- Australia (4):
  - St Vincent's Centre for Applied Medical Research /ID# 249843, Darlinghurst, New South Wales
  - Southern Neurology - Kogarah /ID# 249098, Kogarah, New South Wales
  - Box Hill Hospital /ID# 249095, Box Hill, Victoria
  - Australian Alzheimer's Res Fou /ID# 249097, Nedlands, Western Australia
- Germany (2):
  - Universitaetsklinikum des Saarlandes /ID# 248077, Homburg, Saarland
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 248078, Berlin
- Japan (9):
  - NHO Hiroshima-Nishi Medical center /ID# 256947, Otake-shi, Hiroshima
  - Duplicate_Kawashima Neurology Clinic /ID# 253561, Fujisawa-shi, Kanagawa
  - Shonan Kamakura General Hospital /ID# 256664, Kamakura-shi, Kanagawa
  - Teikyo University Mizonokuchi Hospital /ID# 253259, Kawasaki, Kanagawa
  - Nara Medical University Hospital /ID# 252564, Kashihara-shi, Nara
  - NHO Niigata National Hospital /ID# 254207, Kashiwazaki-shi, Niigata
  - Oita University Hospital /ID# 253679, Yufu, Oita Prefecture
  - Hizen Psychiatric Center /ID# 252363, Kanzaki-gun, Saga-ken
  - Juntendo University Hospital /ID# 252373, Bunkyo-ku, Tokyo
- CGM Research Trust /ID# 249439, Christchurch Central, New Zealand
- Spain (6):
  - Hospital Universitari General de Catalunya /ID# 249100, Sant Cugat del Vallès, Barcelona
  - Hospital Universitari Mútua Terrassa /ID# 248448, Terrassa, Barcelona
  - Hospital Universitario Marques de Valdecilla /ID# 248454, Santander, Cantabria
  - Clinica Universidad de Navarra - Pamplona /ID# 248415, Pamplona, Navarre
  - Hospital Internacional Ruber - Grupo Quiron Salud /ID# 248856, Madrid
  - Hospital Universitario de Salamanca /ID# 249101, Salamanca
- United Kingdom (5):
  - NeuroClin Limited(Previously Glasgow Memory Clinic) /ID# 249787, Motherwell, Lanarkshire
  - Re:Cognition Health Birmingham /ID# 249796, Birmingham
  - Re:Cognition Health Bristol /ID# 249795, Bristol
  - St Pancras Clinical Research /ID# 249006, London
  - Re:Cognition Health - London /ID# 249005, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-515

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo for ABBV-552 once daily (QD) for 12 weeks.
- ABBV-552: 1 mg: Participants received 1 mg of ABBV-552 QD for 12 weeks.
- ABBV-552: 5 mg; ABBV-552: 15 mg: Participants received 5 mg of ABBV-552 QD for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | ABBV-552: 1 mg | ABBV-552: 5 mg | ABBV-552: 15 mg
Started | 66 | 65 | 66 | 66
mITT Population (Modified Intend-to-Treat (mITT) Population included all randomized subjects who received at least 1 capsule of study drug and had at least 1 postbaseline ADAS-Cog 14 score.) | 65 | 63 | 64 | 63
Completed | 63 | 61 | 61 | 60
Not Completed | 3 | 4 | 5 | 6
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 4
Not completed — Other | 0 | 1 | 2 | 1
Not completed — Randomized but Not Treated | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population includes participants who received at least 1 dose of study drug and were grouped according to treatment actually received the majority of the time, defined based on the number of days each treatment was received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ABBV-552: 1 mg | ABBV-552: 5 mg | ABBV-552: 15 mg | Total
Number analyzed (Participants) | 66 | 65 | 65 | 66 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (9.19) | 73.5 (7.33) | 73.2 (7.78) | 73.1 (7.60) | 73.1 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 40 | 43 | 33 | 146
  Male | 36 | 25 | 22 | 33 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 25 | 27 | 22 | 94
  Not Hispanic or Latino | 46 | 40 | 38 | 44 | 168
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 6 | 3 | 7 | 10 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 7 | 7 | 27
  White | 52 | 55 | 51 | 47 | 205
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
ADAS-Cog 14 Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog 14) Score was designed to assess the cognitive impairments most common in AD. It includes the original 11 items from the ADAS-Cog-11 and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in mild cognitive impairment (MCI) patients. The Total Score of the ADAS-Cog-14 ranges from 0 to 90, with a higher score representing greater impairment. Population: Includes mITT participants with data available for analysis.
  units on a scale
    number analyzed (Participants) | 64 | 63 | 64 | 63 | 254
    (all) | 24.10 (8.260) | 22.99 (8.573) | 23.24 (7.780) | 23.82 (8.273) | 23.54 (8.188)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog 14) Score at Week 12
Description: The ADAS-Cog was designed to assess the cognitive impairments most common in AD. The ADAS-Cog-14 includes the original 11 items from the ADAS-Cog-11 [1. Spoken language ability, 2. Comprehension of spoken language, 3. Recall of test instructions, 4. Word-findings difficulty in spontaneous speech, 5. Following commands, 6. Naming objects and fingers, 7. Constructional praxis, 8. Ideational praxis, 9. Orientation, 10. Word-recall task, 11. Word-recognition task] and includes 3 additional tasks [12. Number cancellation task, 13. Delayed word recall task, 14. Executive functioning], for increased sensitivity in mild cognitive impairment (MCI) patients. The Total Score of the ADAS-Cog-14 ranges from 0 to 90, with a higher score representing greater impairment.
Time Frame: Week 12
Population: mITT population includes participants who received at least 1 dose of study drug, have at least 1 post baseline assessment of ADAS-Cog 14, and have data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABBV-552: 1 mg | ABBV-552: 5 mg | ABBV-552: 15 mg
Number analyzed (Participants) | 58 | 56 | 58 | 59
score on a scale | -1.26 (0.660) | -1.28 (0.668) | -1.68 (0.658) | -1.01 (0.655)
Statistical Analysis 1: Comparison: Placebo vs ABBV-552: 1 mg; Test type: Superiority; p = 0.9819, Mixed-effect Model Repeated Measurement; LS Mean of Difference = -0.02, 95% CI 2-sided [-1.87 to 1.83], Standard Error of Mean 0.939
Statistical Analysis 2: Comparison: Placebo vs ABBV-552: 5 mg; Test type: Superiority; p = 0.6545, Mixed-effect Model Repeated Measurement; LS Mean of Difference = -0.42, 95% CI 2-sided [-2.25 to 1.42], Standard Error of Mean 0.931
Statistical Analysis 3: Comparison: Placebo vs ABBV-552: 15 mg; Test type: Superiority; p = 0.7860, Mixed-effect Model Repeated Measurement; LS Mean of Difference = 0.25, 95% CI 2-sided [-1.58 to 2.08], Standard Error of Mean 0.928

ADVERSE EVENTS:
Time Frame: All-cause mortality were reported from enrollment to the end of study, median time on follow up (median time participants were followed) was 116, 116, 115.5, and 114 days for Placebo, ABBV-552:1 mg, 5 mg, and 15 mg arms, respectively. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 30 days after the last dose of study drug; mean duration on study drug was 12 weeks.
Groups:
- ABBV-552: 15 mg: Participants received 15 mg of ABBV-552 QD for 12 weeks.
Arm/Group | Placebo | ABBV-552: 1 mg | ABBV-552: 5 mg | ABBV-552: 15 mg
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/65 | 1/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 3/66 | 3/65 | 2/66 | 2/66
Other Adverse Events (participants affected / at risk) | 15/66 | 16/65 | 19/66 | 20/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=66) | ABBV-552: 1 mg (N=65) | ABBV-552: 5 mg (N=66) | ABBV-552: 15 mg (N=66)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BRUGADA SYNDROME (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=66) | ABBV-552: 1 mg (N=65) | ABBV-552: 5 mg (N=66) | ABBV-552: 15 mg (N=66)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
FATIGUE (General disorders) | 2 (2) | 3 (4) | 2 (3) | 7 (7)
NASOPHARYNGITIS (Infections and infestations) | 2 (3) | 2 (2) | 1 (1) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 4 (5) | 2 (2) | 3 (4)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 5 (7) | 2 (2) | 2 (2) | 2 (2)
DIZZINESS (Nervous system disorders) | 3 (3) | 2 (2) | 4 (4) | 8 (8)
HEADACHE (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT05771428/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT05771428/SAP_001.pdf